CLINICAL TRIAL: NCT04903535
Title: Does a Flashlight Used to Detect Pet Biological Fluids on Human Skin and Other Surfaces Increase Gas Phase Nitric Oxide Levels?
Brief Title: External Nitric Oxide Measurement Through SNO Degradation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Nadzeya V Marozkina, Assistant Research Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10839
Record Dates: First submitted 2021-04-29; First posted 2021-05-26 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-12

CONDITIONS: Healthy; Unconscious
MeSH Terms: conditions — Unconsciousness

STUDY DESIGN:
Intervention Model Description: Healthy Volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Healthy Volunteers (Experimental): Study will enroll to test the assay
  Interventions: Device: Alonefire SV003 10W 365nm UV Flashlight

INTERVENTIONS:
Device: Alonefire SV003 10W 365nm UV Flashlight — Investigator will use a Nitric Oxide Analyzer while attached to a small suction port on the subject's ear lobe to be tested for Nitric Oxide. After getting the baseline assay, the investigator will shine a low-intensity UV Flashlight (Alonefire SV003 10W 365nm UV Flashlight) at the ear lobe for 10 seconds, repeated three times at 20 second intervals, to determine if there is photobleaching. Then the assay will then be performed on the opposite ear lobe. Fifteen minutes after the third UV flashlight exposure, the investigator will collect air from the subject's ear during photolysis into a 20mL glass syringe (once from each ear). Fifteen minutes after the third UV flashlight exposure, the investigator will collect air from the subject's ear during photolysis into a 20mL glass syringe (once from each ear). The subject and the investigator will wear UV goggles during the experiment.

SUMMARY:
In this study, we aim to explore the feasibility of a novel, noninvasive SNO assay to acquire physiological SNO quantification from various parts of the human body and test this new method of analysis. This study aims to help with the currently cumbersome and invasive procedures used to measure SNOs in the body. The proposed activities do not unnecessarily duplicate previous experiments.

DETAILED DESCRIPTION:
S-nitrosylation is the covalent attachment of a nitric oxide group to cystine thiol within a protein to form an S-nitrosothiol (SNO); it has diverse regulatory roles in all mammalian cells and thus operates as a fundamental mechanism for cellular signaling and accounts for a large part of nitric oxide activity. Though SNOs are relevant to many biological disciplines like neuronal, muscular, respiratory, and cardiovascular biology, currently there is no way to measure SNOs that is both easy to use in a clinical setting and accurate in detecting low concentrations; detection is challenging due to the labile nature of the molecules. Low or high concentrations of these molecules could be vital indicators of incoming dangerous issues in the body. A system to easily and accurately measure SNOs could prove useful in preventative treatments. Ultra Violet (UV) light can break SNOs and can be used to measure nitric oxide release, but this method is not fully developed and further research is needed on the potential effect for UV to measure nitric oxide release.

ELIGIBILITY:
Inclusion Criteria

* Adult males or females age ≥ 1 day and ≤ 75 years at time of enrollment

Exclusion Criteria

* Subjects meeting the following criteria will be excluded:
* Smokers.
* Any chronic skin conditions.
* Pregnant.
* Subjects that are unable or unwilling to cooperate with specimen collection.
* Subjects with diagnosis of any medical condition that in the investigator's opinion would make them unsuitable for study participation.
* (for subjects ≥ 18) Subjects that lack the capacity to consent for themselves.

Ages: 1 Day to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Nitric Oxide during UV light exposure | 30 minutes
  NO evolved during UV light exposure from the human ear lobe, hand or forehead.

CONTACTS AND LOCATIONS:
Overall Officials: Nadzeya Marozkina, PhD, MD, Principal Investigator — Indiana University School of Medicine
Locations (2):
- United States (2):
  - Riley Hospital for Children, Indianapolis, Indiana
  - Wells Center for Pediatric Research, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marozkina NV, Gaston B. Nitrogen chemistry and lung physiology. Annu Rev Physiol. 2015;77:431-52. doi: 10.1146/annurev-physiol-021113-170352. PMID 25668023
- [Background] Straub AC, Lohman AW, Billaud M, Johnstone SR, Dwyer ST, Lee MY, Bortz PS, Best AK, Columbus L, Gaston B, Isakson BE. Endothelial cell expression of haemoglobin alpha regulates nitric oxide signalling. Nature. 2012 Nov 15;491(7424):473-7. doi: 10.1038/nature11626. Epub 2012 Oct 31. PMID 23123858
- [Background] Marozkina NV, Gaston B. S-Nitrosylation signaling regulates cellular protein interactions. Biochim Biophys Acta. 2012 Jun;1820(6):722-9. doi: 10.1016/j.bbagen.2011.06.017. Epub 2011 Jun 24. PMID 21745537
- [Background] Palmer LA, Gaston B. S-nitrosothiol assays that avoid the use of iodine. Methods Enzymol. 2008;440:157-76. doi: 10.1016/S0076-6879(07)00809-9. PMID 18423216